CLINICAL TRIAL: NCT01032499
Title: Multicenter Clinical Study,Phase III, Prospective, Randomized, Open and Comparative to Measure Tolerability and Efficacy of Taro Elixir on the Evolution Treatment of Acne Vulgaris II and III Degree or of Furunculosis Compared With Oxytetracycline
Brief Title: Open and Comparative Study to Measure Tolerability and Efficacy of Taro Elixir
Acronym: E01GOU-INH0109
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorios Goulart S.A. (Industry)
Responsible Party: Voltaire Gominho de Oliveira, Laboratorios Goulart S.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E01-GOU-INH-01-09
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-12

CONDITIONS: Acne Vulgaris II or III Degree; Boils
Keywords: Acne Vulgaris; Boil; Taro Elixir
MeSH Terms: conditions — Furunculosis; Acne Vulgaris | interventions — Oxytetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxytetracycline (Active Comparator)
  Interventions: Drug: oxytetracycline, taro elixir
- Taro Elixir (Experimental): Taken orally one tablespoon (15 mL) of Taro Elixir 3 times daily for breakfast, lunch and dinner.
  Interventions: Drug: Taro Elixir

INTERVENTIONS:
Drug: oxytetracycline, taro elixir — comparison of treatment efficacy between oxytetracycline and taro elixir
  Arms: oxytetracycline
Drug: Taro Elixir — Taken orally one tablespoon (15 mL) of Taro Elixir 3 times daily for breakfast, lunch and dinner.
  Arms: Taro Elixir

SUMMARY:
To measure the efficacy of Taro Elixir compare with Oxytetracycline in the treatment of boils or acne.

ELIGIBILITY:
Inclusion Criteria:

* Both of gender patient, older than 14 years;
* Patient with boils or acne vulgaris II or III degree;
* The score must be at least than 4, for 2 or more question of VAS (visual analog scale);
* Patient that have been used an effective contraceptive method in the last 3 months, including sexual abstinence and that keep using that method during the study until a month after;
* Patient that have been accepted to participate of the study and signed the Informed Consent or in case of younger than 18 years, the responsable must read and sign the Informed Consent.
* Patient that have been accepted to meet all the visits stipulated at the protocol, whenever the investigator request in .

Exclusion Criteria:

* Patient of female gender that has been pregnant, breastfeeding or that has not been use a safe contraceptive method (oral contraceptives or barrier methods). Sexual abstinence will be accept if the investigator think that it is relevant.
* Patient that has been use antiandrogens (cyproterone, finasteride, flutamide, tamoxifen, spironolactone);
* Patient with acne I or IV degree;
* Patient that has been receive some treatment for acne as antibiotics, corticosteroid or any medicine that can maybe interfere in the study results: a month for systemic treatment or two weeks for topic treatment, before inclusion or during the study;
* Patient that received treatment with oral retinoids within 6 months before the inclusion and during the study;
* Patient that had a known decompensated diabetes history;
* Patient with immunodeficiency and liver, renal, cardiac, digestive, metabolic, endocrinological, hematological, neurological or psychiatric disorders, evaluated through anamnesis by the investigator, tha can maybe interfere on the study evaluation. Even the patient with facial dermatoses such as psoriasis, acne rosacea, allergic dermatitis, skin infections caused by fungi, bacteria and viruses;
* Patient with alcoholism history, illicit drugs use, psychological ou emotional problems that can maybe void the Informed Consent or limit the capacity of the patient follow the protocol requirements ;
* Patient hypersensitive to any one of the medicine components;
* Patient that have been used any drug under search, 3 months before the visit number one.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Measure the efficacy in the treatment of boils or acne vulgaris II and III degree with taro elixir compared with Oxytetracycline. | 90 days

SECONDARY OUTCOMES:
Measure the tolerability in the treatment evolution of boils or acne vulgaris II and III with taro elixir compare with Oxytetracycline. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Machado, Principal Investigator — Faculdade de Medicina do ABC; Andrea Gerbase, Principal Investigator — Alergoclínica - Centro de Alergia e dermatologia; Denise Steiner, Principal Investigator — Policlínica Mogi das Cruzes; Jussara Marin, Principal Investigator — Alergoclínica - Centro de alergia e dermatologia
Locations (3):
- Brazil (3):
  - Policlínica de Mogi das Cruzes, Mogi das Cruzes, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Alergoclínica - Centro de alergia e dermatologia, São Paulo, São Paulo